CLINICAL TRIAL: NCT04502199
Title: Dysautonomic Signs Among MECP2boys
Brief Title: Dysautonomic Phenotype in Male Patients With MECP2 Mutation
Acronym: MECP2BOYS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: MECP2BOYS (29BRC20.0182)
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: MECP2-Related Severe Neonatal Encephalopathy; Dysautonomia; Masculinity
MeSH Terms: conditions — Encephalopathy, Neonatal Severe, Due To Mecp2 Mutations; Autonomic Nervous System Diseases; Masculinity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional study — observational study

SUMMARY:
Dysautonomic signs are well known among girls with a Rett Syndrom. Rett syndrom is caused by a MECP2 mutation in 95% of cases. We want to search dysautonomic signs among boys with a MECP2 mutations because they are less studied than the girls and they have more varied phenotypes.

DETAILED DESCRIPTION:
First, we will launch a national call for participation in all the genetics departments in France to research boys with a missense or a non-sens mutation in the MECP2 gene. Our inclusion criteria is : less than 16 years old or dead before 16 years old patients of masculin sex with a missense or non-sens mutation in the MECP2 gene. Exclusion criteria is : patient under judicial protection or participation refusal by one of the legal guardian. Inclusion will take place in August 2020.

We had conceived an excel spreadsheet (2007 version) to collect all the datas needed with general data such as age, genetic mutation with the HGVS nomenclature using the NM_001110792.2, familial and personal history, mensurations, dysmorphic signs. To search dysautonomic signs, we used a system approach. We will look for neurological signs : abnormal movements, sleep disturbance, cardiologic signs :abnormal bradycardia or tachycardia, hypotension, rythms anomalies, respiratory signs : respiratory irregularities, apnea, hyperpnea , digestive signs : gastrooesophagal reflux, constipation, diarrhea, vomiting or subocclusif episodes, thermoregulation signs : abnormal hypo or hyperthermia, excessive sweating. Each time a dysautonomic sign will be reported in a letter of a patient, we will demand this sign to be objectived by a complementary exam, or by a precise device during an hospitalisation : electoencephalogram (EEG), polysomnography (PSG), Electrocardiogram (ECG), holter-ECG, digestive fibroscopies, scoped surveillance.

If we have a positive response, we will contact the main caregiver of the patient who can be a neurologist or a geneticist and will provid him a spreadsheet and an explanatory sheet. We will ask of him a systematic review of all the letters of the patient including letters of hospitalisation, of the specialists, complementary exams. A non-opposition letter will be sent to him in a way he can send it to the legal guardians of the children : a non-opposition of 15 days will be requested. Then, the filled spreadsheet will be sent back to the center of inclusion in Brest through a securised mailbox. Data will be kept on a secure database with a password.

Our primary endpoint is the presence of at least one dysautonomic sign. We intend to include between 10 and 20 patients in this multicentric study. To analyse our results, we will use a descriptive approach.

This protocole was validated by the Ethic Comitee of Brest in june 18, 2020

ELIGIBILITY:
Inclusion Criteria:less than 16 years old or dead before 16 years old patients of masculin sex with a missense or non-sens mutation in the MECP2 gene -

Exclusion Criteria:patient under judicial protection or participation refusal by one of the legal guardian

-

Max Age: 16 Years | Sex: Male
Age Groups: Child
Gender Based: Yes
Study Population: less than 16 years old or dead before 16 years old patients of masculin sex with a missense or non-sens mutation in the MECP2 gene
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2021-01-13 (Estimated); Study Completion 2021-01-13 (Estimated)

PRIMARY OUTCOMES:
presence of at least one dysautonomic sign | one month

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU de Besançon, Besançon
  - CHRU de Brest, Brest
  - CHRU de Lille, Lille
  - Hospices Civiles de Lyon, Lyon
  - Hôpital de la Timone, Marseille
  - CHU de NIMES, Nîmes
  - Hôpital Robert Debre, Paris

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning six months and ending five years following the end study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.